CLINICAL TRIAL: NCT02434302
Title: Characteristics and Outcomes of Childhood Moyamoya in the UK
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13NR31
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Moyamoya
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study to ascertain the number of children with moyamoya in the UK, their presenting features, clinical course and outcomes.

DETAILED DESCRIPTION:
The study ahs 3 components:

1. Patient identification via the British Paediatric Surveillance Unit, and the 21 collaborating centres
2. Record review/patient interview to determine clinical features & outcomes
3. Centralised review of imaging data to ascertain radiological phenotypes

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of moyamoya

Exclusion Criteria:

* Refuse consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (0-18y) with moyamoya in the UK over study period (2014-2016 August)
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of children with moyamoya in UK | 2 years

SECONDARY OUTCOMES:
clinical features & outcomes of childhood moyamoya | 2 years
radioplogical features of childhood Moyamoya | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: vijeya ganesan, MB ChB MD, Principal Investigator — UCL Institute of Child Health
Locations (1):
- Great Ormond Street Hospital for CHidlren NHS Foundation Trust, London, United Kingdom